CLINICAL TRIAL: NCT04917588
Title: A Prospective, Open-label, Multicentre, Randomized Study to Evaluate the Effectiveness, Safety and Long Term Safety of Saypha® FILLER Lidocaine for Lip Augmentation
Brief Title: Study to Evaluate the Effectiveness, Safety and Long Term Safety of Saypha® FILLER Lidocaine for Lip Augmentation
Acronym: SayLip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPH-101-201479
Record Dates: First submitted 2021-05-26; First posted 2021-06-08 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2022-05

CONDITIONS: Abnormal Lip
Keywords: Moderate to Severe Lip Volume Deficit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saypha® FILLER HQ (Experimental): Eligible subjects will undergo bilateral lip augmentation treatments with Saypha® FILLER Lidocaine manufactured in the Croma Pharma HQ Facility in order to correct moderate to severe deficiency of lip volume.
  The treatment will be administered at the Baseline visit (Day 0).
  Interventions: Combination Product: Saypha® FILLER Lidocaine (HQ)
- Saypha® FILLER C1 (Active Comparator): Eligible subjects will undergo bilateral lip augmentation treatments with Saypha® FILLER Lidocaine manufactured in the Croma Pharma C1 Facility in order to correct moderate to severe deficiency of lip volume.
  The treatment will be administered at the Baseline visit (Day 0).
  Interventions: Combination Product: Saypha® FILLER Lidocaine (C1)

INTERVENTIONS:
Combination Product: Saypha® FILLER Lidocaine (HQ) — Saypha® FILLER Lidocaine is administered by injection into the lips. The volume applied depends on the size of the area which requires correction and will be selected by the investigator. A maximum volume of 2 mL for both lips in total (i.e., for upper plus lower lip) including touch up might be needed per treatment but the treatment should not exceed 10 mL in total per treatment or 20 mL per year.
  Arms: Saypha® FILLER HQ
Combination Product: Saypha® FILLER Lidocaine (C1) — Saypha® FILLER Lidocaine is administered by injection into the lips. The volume applied depends on the size of the area which requires correction and will be selected by the investigator. A maximum volume of 2 mL for both lips in total (i.e., for upper plus lower lip) including touch up might be needed per treatment but the treatment should not exceed 10 mL in total per treatment or 20 mL per year.
  Arms: Saypha® FILLER C1

SUMMARY:
This is a prospective, open-label, multicentre, randomized study conducted to evaluate the effectiveness, safety and long-term safety of Saypha® FILLER Lidocaine for lip augmentation.

DETAILED DESCRIPTION:
Following informed consent and screening, eligible subjects with moderate to severe deficiency of lip volume will be randomized to receive Saypha® FILLER Lidocaine from 1 of 2 manufacturing sites. The device will be injected into the submucosa of the lips, and subjects will return for follow-up assessments at Week 3, 6, 26, 52 and optional at Week 76 after the treatment.

A Touch-up treatment may be done at Week 3, if deemed appropriate by the investigator. The performance of the investigational device will be evaluated by the investigator by assessing severity using the LFS, Lip Fullness Scale, at Week 6, 26, 52 after the treatment and optional at Week 76 and in comparison to Day 0. The upper and lower lip will be graded separately.

Telephone visits will be performed approximately 24 hours post-administration to monitor possible adverse events. In case any adverse events are reported during the telephone visits an unscheduled visit should be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female or male subjects 18 years of age at Screening/Baseline visit (Visit 1)
2. Presence of approximately symmetrical "very thin" lips (minimal red lip shows) to "moderately thick" lips (moderate red lip shows) as assessed with the LFS (severity grade of 1 to 3 on both lips) as determined by the investigator at Visit 1
3. For females of childbearing potential only: negative urine pregnancy test at Visit 1, and must agree to use an highly effective method of contraception for the duration of the clinical investigation
4. Healthy skin in the treatment area and free of diseases that could interfere in evaluation of treatment
5. Willingness to abstain from any cosmetic or surgical procedures in the treatment area for the duration of the clinical investigation
6. Willingness to take part in this clinical investigation documented by a personally signed/dated informed consent.

Exclusion Criteria:

1. Pregnancy, lactation, planned pregnancy or unwillingness to use contraception at any time during the study (for women of child-bearing potential only)
2. History of mental disorders or emotional instability
3. History of allergic reaction or hypersensitivity to hyaluronic acid, lidocaine or any amide-based anaesthetic
4. Prior surgery, scars or tattoo to the upper or lower lip or lip line; surgery and tattooing are prohibited until end of clinical investigation
5. Tooth gap, overbite, beard longer three-day beard, or excessive facial hair that could interfere in evaluation of treatment as judged by the investigator
6. Presence of any abnormal lip structure, such as a scar or lump or severe lip asymmetry, as judged by the investigator
7. Previous tissue augmenting therapy in the lip area (including lips, oral commissures, nasolabial folds, marionette and perioral lines) with HA or collagen filler, or laser treatment, chemical peeling, dermabrasion or mesotherapy within 12 months before Visit 1 and until end of clinical investigation
8. Previous permanent implant or treatment with non-HA or non-collagen filler in the lip area (including lips, oral commissures, nasolabial folds, marionette and perioral lines) and until end of the investigation
9. Previous toxin treatment in the lip area (including lips, oral commissures, nasolabial folds, marionette and perioral lines) within 9 months before Visit 1 and until end of clinical investigation
10. Presence of cutaneous lesions, inflammatory and/or infectious processes (e.g. acne, herpes, etc.) or proliferative lesions in the treatment area
11. Known human immune deficiency virus-positive individuals
12. History of allergies against aesthetic filling products and recurrent (3 times a year) herpes simplex in the treated area
13. Tendency to hypertrophic scars, keloid formation and/or pigmentation disorders
14. History or presence of any autoimmune or connective tissue disease, or current treatment with immune therapy
15. Uncontrolled systemic diseases (such as diabetes mellitus)
16. Use of anticoagulant, antiplatelet or thrombolytic medication (e.g. acetylsalicylic acid) from 10 days pre- to three days post IMD injections
17. Planned dental/oral surgery or modification (bridge-work, implants) within two weeks prior to initial IMD injection and to a minimum of four weeks post IMD injections
18. Any medical condition which, in the investigator's opinion, prohibits the inclusion in the study
19. Current or previous (within 30 days of enrolment) treatment with another investigational drug and/or medical device or participation in another clinical study
20. Previous enrolment in this clinical investigation
21. Any dependent relationship of the subject with the investigator, investigation site or Sponsor (e.g. employees or relatives)
22. Subjects whose participation in clinical trials is prohibited by the Austrian Medical Devices Act (e.g., persons with a legal custodian appointed due to mental disability, prisoners, soldiers and other members of the armed forces, civil servants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Medizinisch Aesthetisches Zentrum Wien, Vienna
  - YUVELL - Home of Aesthetics, Vienna
  - PW-Privatklinik Waehring GmbH, Vienna

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screened patients: N=121; Screening failures: N=7; Patients enrolled = Patients Treated with IMD: N= 114
Groups:
- Saypha® FILLER HQ: Eligible subjects will undergo bilateral lip augmentation treatments with Saypha® FILLER Lidocaine manufactured in the Croma Pharma HQ Facility in order to correct moderate to severe deficiency of lip volume.
  The treatment will be administered at the Baseline visit (Day 0).
  Saypha® FILLER Lidocaine (HQ): Saypha® FILLER Lidocaine is administered by injection into the lips. The volume applied depends on the size of the area which requires correction and will be selected by the investigator. A maximum volume of 2 mL for both lips in total (i.e., for upper plus lower lip) including touch up might be needed per treatment but the treatment should not exceed 10 mL in total per treatment or 20 mL per year.
- Saypha® FILLER C1: Eligible subjects will undergo bilateral lip augmentation treatments with Saypha® FILLER Lidocaine manufactured in the Croma Pharma C1 Facility in order to correct moderate to severe deficiency of lip volume.
  The treatment will be administered at the Baseline visit (Day 0).
  Saypha® FILLER Lidocaine (C1): Saypha® FILLER Lidocaine is administered by injection into the lips. The volume applied depends on the size of the area which requires correction and will be selected by the investigator. A maximum volume of 2 mL for both lips in total (i.e., for upper plus lower lip) including touch up might be needed per treatment but the treatment should not exceed 10 mL in total per treatment or 20 mL per year.
Period: Overall Study
Arm/Group | Saypha® FILLER HQ | Saypha® FILLER C1
Started | 57 | 57
Completed | 50 | 51
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Population: Population considered for this analysis is the Full Analysis Set (FAS) which comprises all subjects who received at least 1 administration of the IMD and who had at least 1 post-treatment evaluation of the LFS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saypha® FILLER HQ | Saypha® FILLER C1 | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (13.78) | 44.4 (16.22) | 43.2 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 57 | 114
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 57 | 57 | 114
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 57 | 57 | 114
Smoking habit [Count of Participants; unit: Participants] — Smoking habit: Former smoker: greater than 3 months since smoking cessation; Current smoker: less than 3 months since smoking cessation
  Participants
    current | 21 | 22 | 43
    former | 4 | 4 | 8
    never smoked | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate in Lip Volume Improvement
Description: The proportion of subjects ('responders') with the lip volume improved by ≥1 point versus baseline value at 6 weeks after initial treatment based on the investigator live assessment using the validated Lip Fullness Scale (LFS). Lip Fullness Scale (LFS) is a validated 5-point rating scale,that evaluates the Lip Volume Deficiency ranging from Grade 1 (minimal volume) to Grade 5 (very significant volume): In this case, the bigger the number, the better.
Time Frame: Week 6
Population: Population considered for this analysis is the Full Analysis Set (FAS) which comprises all subjects who received at least 1 administration of the IMD and who had at least 1 post-treatment evaluation of the LFS.
  Individual LFS grades per visit are calculated separately for the upper and the lower lip.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Population (Saypha® FILLER HQ + Saypha® FILLER C1): Total eligible subjects that had bilateral lip augmentation treatments with both Saypha® FILLER Lidocaine manufactured in the Croma Pharma C1 Facility and with Saypha® FILLER Lidocaine manufactured in the Croma Pharma in HQ facility.
Arm/Group | Saypha® FILLER HQ | Saypha® FILLER C1 | Overall Population (Saypha® FILLER HQ + Saypha® FILLER C1)
Number analyzed (Participants) | 56 | 54 | 110
Participants
  lower lip responders | 55 | 52 | 107
  upper lip responders | 53 | 53 | 106

2. Secondary Outcome: Percentage of Responders Based on the Investigator Live Assessment
Description: The percentage of responders (with the Lip Volume Improved by >=1 Point Versus Baseline Value,) based on the investigator live assessment at 6, 12 and optional 18 months after the initial treatment using the validated LFS.
  Lip Fullness Scale (LFS) is a validated 5-point rating scale,that evaluates the Lip Volume Deficiency ranging from Grade 1 (minimal volume) to Grade 5 (very significant volume): In this case, the bigger the number, the better.
Time Frame: 6, 12 and optional 18 months
Population: FAS (defined in the Analyis Population description of the primary outcome measure) was considered for the analysis of the secondary endpoints.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Population ( Saypha® FILLER HQ + Saypha® FILLER C1): Total eligible subjects that had bilateral lip augmentation treatments with both Saypha® FILLER Lidocaine manufactured in the Croma Pharma C1 Facility and with Saypha® FILLER Lidocaine manufactured in the Croma Pharma in HQ facility.
Arm/Group | Saypha® FILLER HQ | Saypha® FILLER C1 | Overall Population ( Saypha® FILLER HQ + Saypha® FILLER C1)
Number analyzed (Participants) | 56 | 54 | 110
Participants
  Month 6 Lower Lips | 48 | 50 | 98
  Month 6 Upper Lips | 49 | 50 | 99
  Month 12 Lower Lips | 41 | 36 | 77
  Month 12 Upper Lips | 38 | 36 | 74
  Month 18 Lower Lips | 28 | 23 | 51
  Month 18 Upper Lips | 24 | 19 | 43

3. Secondary Outcome: Percentage of Responders Based on the Independent Photographic Reviewer´s Assessments
Description: The percentage of responders based on the independent photographic reviewer´s assessments at Week 6, Month 6, 12 and optional Month 18 after initial treatment, based on photographs and using the validated LFS (compared to Baseline). Lip Fullness Scale (LFS) is a validated 5-point rating scale,that evaluates the Lip Volume Deficiency ranging from Grade 1 (minimal), Grade 2 (slight), Grade 3 (moderately thick), Grade 4 (thick), to Grade 5 (very significant): In this case, the bigger the number, the better.
Time Frame: Week 6, Month 6, 12 and optional Month 18
Population: FAS - see primary endopoint for FAS definition
Measure: Count of Participants; unit: Participants
Arm/Group | Saypha® FILLER HQ | Saypha® FILLER C1 | Overall Population ( Saypha® FILLER HQ + Saypha® FILLER C1)
Number analyzed (Participants) | 56 | 54 | 110
Participants
  Week 6 - Lower Lip | 25 | 30 | 55
  Week 6 - Upper Lip | 17 | 25 | 42
  Month 6 - Lower Lip | 20 | 19 | 39
  Month 6 - Upper Lip | 15 | 24 | 39
  Month 12 - Lower Lip | 20 | 15 | 35
  Month 12 - Upper Lip | 20 | 26 | 46
  Month 18 - Lower Lip | 15 | 16 | 31
  Month 18 - Upper Lip | 13 | 21 | 34

4. Secondary Outcome: Percentage of Subjects With an Improvement Based on the Investigator Assessment Using GAIS
Description: The percentage of subjects with an improvement relative to baseline photographs, (subjects who have been rated as "very much improved" or "much improved" or "improved"), based on the investigator assessment at Week 6, Month 6, 12 and optional Month 18 after initial treatment using the 5-point GAIS.
Time Frame: Week 6, Month 6, 12 and optional Month 18
Population: FAS - Please see primary endpoint for definition
Measure: Count of Participants; unit: Participants
Arm/Group | Saypha® FILLER HQ | Saypha® FILLER C1 | Overall Population ( Saypha® FILLER HQ + Saypha® FILLER C1)
Number analyzed (Participants) | 56 | 54 | 110
Participants
  Week 6 -Lower Lip | 56 | 54 | 110
  Week 6 - Upper Lip | 56 | 54 | 110
  Month 6 - Lower Lip | 53 | 53 | 106
  Month 6 - Upper Lip | 53 | 53 | 106
  Month 12- Lower Lip | 44 | 41 | 85
  Month 12 - Upper Lip | 44 | 40 | 84
  Month 18 - Lower Lip | 30 | 26 | 56
  Month 18 -Upper Lip | 30 | 21 | 51

5. Secondary Outcome: Percentage of Subjects With an Improvement Based on Subject Assessment Using GAIS
Description: The percentage of subjects with an improvement relative to baseline photographs (subjects who have been rated as "very much improved" or "much improved" or "improved"), based on subject assessment at Week 6, Month 6, 12 and optional Month 18 after initial treatment, using the 5-point GAIS with results ranging from 1 to 5 with lower numbers indicating better improvement
Time Frame: Week 6, Month 6, 12 and optional Month 18
Population: FAS - please see primary endpoint description
Measure: Count of Participants; unit: Participants
Arm/Group | Saypha® FILLER HQ | Saypha® FILLER C1 | Overall Population ( Saypha® FILLER HQ + Saypha® FILLER C1)
Number analyzed (Participants) | 56 | 54 | 110
Participants
  Week 6 - lower lips | 55 | 54 | 109
  Week 6 - upper lips | 56 | 54 | 110
  Month 6 - Lower Lips | 51 | 53 | 104
  Month 6 - Upper Lips | 53 | 53 | 106
  Month 12 - Lower Lips | 45 | 44 | 89
  Month 12 - Upper Lips | 44 | 44 | 88
  Month 18 - Lower Lips | 37 | 34 | 71
  Month 18 - Upper Lips | 34 | 35 | 69

6. Secondary Outcome: Subject Satisfaction Using Face-Q Questionnaire
Description: The extent of subject´s satisfaction with overall outcome of the treatment, at Week 6, Month 6, 12 and optional Month 18 after initial treatment, assessed by the subject using the Face-Q TM Questionnaire. The FACE-Q Satisfaction with Outcome scale is a patient-reported outcome measure designed to assess a patient's satisfaction with the results of a facial aesthetic procedure. This scale comprises six items, each with four response options: "definitely agree," "somewhat agree," "somewhat disagree," and "definitely disagree." The raw summed scale score is converted to a score from 0 to 100 by using the respective Conversion Tables available from Face Q authors. Higher scores reflect a better outcome (i.e., 0 (worst) to 100 (best)).
Time Frame: Week 6, Month 6, 12 and optional Month 18
Population: The population considered for this analysis comprises all subjects who received at least 1 administration of the Investigational Medical Device, who had at least 1 post-treatment evaluation using the Lip Fullness Scale and who have Face-Q measurements available for the respective timepoints. In the protocol and statistical analysis plan, the analysis for this outcome measure was planned only for the overall population and not for the randomized subgroups Saypha® FILLER HQ and Saypha® FILLER C1.
Measure: Mean (Standard Deviation); unit: score on Face Q questionnaire
Arm/Group | Overall Population ( Saypha® FILLER HQ + Saypha® FILLER C1)
Number analyzed (Participants) | 110
score on Face Q questionnaire
  Week 6 | 85.8 (17.88)
  Month 6: number analyzed (Participants) | 108
  Month 6 | 80.0 (20.61)
  Month 12: number analyzed (Participants) | 106
  Month 12 | 71.7 (25.53)
  Month 18: number analyzed (Participants) | 81
  Month 18 | 78.3 (25.76)

7. Secondary Outcome: Subject Satisfaction Using Face-Q TM Questionnaire "Satisfaction With Lips"
Description: The extent of subject's satisfaction with augmentation of lips, at Week 6, Month 6, 12 and optional Month 18 after initial treatment, assessed by the subject using the Face-Q TM Questionnaire "Satisfaction with Lips", a 6-items Aesthetic Appearance Questionnaire with 5 pre-defined answer options between "very satisfied" and "very dissatisfied".
  The extent of subject´s satisfaction with overall outcome of the treatment, at Week 6, Month 6, 12 and optional Month 18 after initial treatment, assessed by the subject using the Face-Q.
  The raw summed scale score is converted to a score from 0 to 100 by using the respective Conversion Tables available from Face Q authors. Higher scores reflect a better outcome (i.e., 0 (worst) to 100 (best)).
Time Frame: Week 6, Month 6, 12 and optional Month 18
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score Face Q questionnaire
Arm/Group | Overall Population ( Saypha® FILLER HQ + Saypha® FILLER C1)
Number analyzed (Participants) | 110
score Face Q questionnaire
  Week 6 | 90.9 (11.96)
  Month 6: number analyzed (Participants) | 108
  Month 6 | 84.9 (17.24)
  Month 12: number analyzed (Participants) | 106
  Month 12 | 76.2 (22.69)
  Month 18: number analyzed (Participants) | 81
  Month 18 | 78.3 (20.45)

8. Secondary Outcome: Subject's Perception of Pain Using the 11-point Numeric Pain Rating Scale
Description: Subject's perception of pain after initial and touch-up treatment with Saypha® FILLER Lidocaine using the 11-point Numeric Pain Rating Scale (NPRS), where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: Day1, Week 3
Population: FAS-please see primary endpoint population definition
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Saypha® FILLER HQ: Eligible subjects that had bilateral lip augmentation treatments with both Saypha® FILLER Lidocaine manufactured in Croma Pharma HQ facility.
- Saypha® FILLER C1: Eligible subjects that had bilateral lip augmentation treatments with Saypha® FILLER Lidocaine manufactured in the Croma Pharma C1 facility.
Arm/Group | Overall Population ( Saypha® FILLER HQ + Saypha® FILLER C1) | Saypha® FILLER HQ | Saypha® FILLER C1
Number analyzed (Participants) | 110 | 56 | 54
score on a scale
  Initial Treatment - Immediately after treatment | 3.3 (1.71) | 3.6 (1.75) | 3.0 (1.62)
  Initial Treatment - 15 min post treatment | 0.5 (0.92) | 0.7 (1.05) | 0.3 (0.73)
  Touch up (Week 3) - Immediately after treatment: number analyzed (Participants) | 54 | 25 | 29
  Touch up (Week 3) - Immediately after treatment | 2.9 (1.48) | 2.7 (1.52) | 3.0 (1.46)
  Touch up (Week 3 ) - 15 min post treatment: number analyzed (Participants) | 54 | 25 | 29
  Touch up (Week 3 ) - 15 min post treatment | 0.4 (0.65) | 0.4 (0.77) | 0.3 (0.53)

9. Secondary Outcome: Percentage of Subjects Demonstrating an Aesthetic Effect
Description: Percentage of subjects demonstrating an aesthetic effect at Week 6, Month 6, 12 and optional Month 18 based on the investigator's life assessment.
  A live assessment of the treated areas was performed and the treated areas compared to the subject's photographs obtained at the Baseline Visit. The presence of the aesthetic effect was recorded as either "Yes" or "No"
Time Frame: Week 6, Month 6, 12 and optional Month 18
Population: The population considered for this analysis comprises all subjects who received at least 1 administration of the Investigational Medical Device and who had at least 1 post-treatment evaluation using the Lip Fullness Scale. In the protocol and statistical analysis plan, the analysis for this outcome measure was planned only for the overall population and not for the randomized subgroups Saypha® FILLER HQ and Saypha® FILLER C1.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Population ( Saypha® FILLER HQ + Saypha® FILLER C1)
Number analyzed (Participants) | 110
Participants
  Week 6 | 110
  Month 6 | 106
  Month 12 | 86
  Month 18 | 59

10. Secondary Outcome: Injection Volume Required
Description: Injection volume (initial and touch-up) required for an optimal augmentation of the lips with Saypha® FILLER Lidocaine.
Time Frame: Day1, Week 3
Population: The population considered for this analysis comprises all subjects who had at least 1 post-treatment evaluation using the Lip Fullness Scale and who received treatment with the Investigational Medical Device at the respective timepoints. In the protocol and statistical analysis plan, the analysis for this outcome measure was planned only for the overall population and not for the randomized subgroups Saypha® FILLER HQ and Saypha® FILLER C1.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Overall Population ( Saypha® FILLER HQ + Saypha® FILLER C1)
Number analyzed (Participants) | 110
ml
  Day 1 - initial treatment -lower lip | 0.79 (0.282)
  Day 1 - Initial Treatment - Upper Lip | 0.80 (0.285)
  Day 1 - initial treatment - both lips | 1.59 (0.516)
  Week 3 - touch up treatment - lower lip: number analyzed (Participants) | 39
  Week 3 - touch up treatment - lower lip | 0.50 (0.298)
  Week 3 - touch up treatment - upper lip: number analyzed (Participants) | 51
  Week 3 - touch up treatment - upper lip | 0.51 (0.305)
  Week 3 - touch up treatment - both lips: number analyzed (Participants) | 54
  Week 3 - touch up treatment - both lips | 0.85 (0.604)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were documented from the time of first IMD application at Baseline visit (Visit 1) throughout the course of the clinical investigation, which means up to 18 months after IMD application.
Description: AEs will be detected at each visit by observation and by asking the subject about the occurrence of AEs. Care should be taken not to introduce bias when eliciting AE information from the subject. Open-ended and non-leading verbal questioning is the preferred method. In addition, the subjects will be instructed to immediately contact the investigator/investigation site in case of occurrence of any untoward event between visits and an unscheduled visit will be performed.
Arm/Group | Saypha® FILLER HQ | Saypha® FILLER C1
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 1/57
Other Adverse Events (participants affected / at risk) | 35/57 | 32/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saypha® FILLER HQ (N=57) | Saypha® FILLER C1 (N=57)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) — Worsening of Depression
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saypha® FILLER HQ (N=57) | Saypha® FILLER C1 (N=57)
Application site pain (General disorders) | 26 (30) | 21 (25) — This event is related with the context of an injection site reaction
Injection Site Bruising (General disorders) | 17 (21) | 16 (22) — Injection site reaction
Injection site swelling (General disorders) | 18 (22) | 16 (22) — Injection site reaction
COVID 19 (Infections and infestations) | 11 (13) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT04917588/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT04917588/SAP_001.pdf